CLINICAL TRIAL: NCT00501956
Title: Randomized Study on the Effect of Intradialytic Parenteral Nutrition in Malnourished Hemodialysis Patients
Brief Title: Intradialytic Parenteral Nutrition in Hemodialysis Patients
Acronym: IDPNHD
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Fresenius Kabi (Industry)
Collaborators: Institute for Clinical Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IDPN 24332
Record Dates: First submitted 2007-07-16; First posted 2007-07-17 (Estimated); Last update posted 2016-03-03 (Estimated); Status verified 2016-03

CONDITIONS: Malnutrition; Complication of Hemodialysis
Keywords: chronic renal replacement therapy; malnutrition anorexia; parenteral nutrition
MeSH Terms: conditions — Malnutrition; Hyperphagia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intradialytic parenteral nutrition (Experimental): Individually compounded intradialytic parenteral nutrition (IDPN) including glucose, amino acids, lipids, L-Carnitine, trace elements and water-soluable vitamins 3x / week over 16 weeks + 12 weeks postinterventional observation.
  Interventions: Drug: Intradialytic Parenteral Nutrition (IDPN)
- Control Group (No Intervention): Observation over 28 weeks (16 + 12 weeks).

INTERVENTIONS:
Drug: Intradialytic Parenteral Nutrition (IDPN) — compounded IDPN, 3 x/week, 16 weeks intervention
  Other Names: Individually compounded parenteral nutrition
  Arms: Intradialytic parenteral nutrition

SUMMARY:
Malnutrition is a major cause of death in chronic hemodialysis patients. Primary treatment of malnutrition in these patients is dietetic counseling, additional enteral nutrition and occasionally drug therapy.

In cases where primary treatment of malnutrition is not effective, intradialytic parenteral nutrition (IDPN)during dialysis therapy may be administered. Using IDPN aminoacids, carbohydrates and fatty acids as well as vitamins and trace elements can be given to the patients.

Effectiveness of IDPN has to be verified.

DETAILED DESCRIPTION:
25% of hemodialysis patients who are treated for more than 5 years suffer from protein malnutrition. 7% have a protein catabolic rate less than 0,6 g/kgBW and day.

The conventional treatment of malnutrition include dietetic counseling, psychologic advice and giving additional oral nutrients.In many cases this kind of therapy is uneffective. If supplementary enteral nutrition is used, the additional intake of water has to be taken into consideration.

IDPN is a mode of treatment by which disadvantages of enteral nutrition and fluid overload of the patients can be avoided.During each dialysis session nutrients can be given and additional water simultaneously can be removed by ultrafiltration.

Some publications have shown that the catabolic state of the patients can be converted into an anabolic state. There are only small randomized studies showing the positive effect of IDPN.

In this german multicenter study malnourished hemodialysis patients are randomized into two groups. One group is treated with IDPN during each dialysis session for 16 weeks followed by 12 weeks of follow-up without IDPN. The control-group does not receive IDPN.

The parameters of metabolism are: Albumin, prealbumin, transferrin, phase angle alpha (bioimpedance), proteincatabolic rate (formal urea kinetics), BMI and subjective global assessment (SGA score).

ELIGIBILITY:
Inclusion Criteria:

* hemodialysis therapy more than 6 months
* three times per week hemodialysis
* albumin < 35 g/l
* prealbumin < 250 mg/l
* phase angle < 4,5°
* SGA score grade B or C
* informed consent

Exclusion Criteria:

* inadequate dialysis (Kt/V < 1,2)
* chemotherapy or radiotherapy
* cardiac pacemaker
* acute bacterial infection
* acute immunological disease
* cancer disease
* severe hepatic insufficiency
* interferon therapy
* HIV disease
* severe diabetes mellitus

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2004-07; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Change in prealbumin levels | 8 weeks

SECONDARY OUTCOMES:
Serum albumin, transferrin, nutritional status | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Helmut Mann, Prof. Dr., Principal Investigator — Interneph e.V, Aachen
Locations (1):
- Interneph e.V. Institute for Applied Nephrology, Aachen, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mitch WE. Malnutrition: a frequent misdiagnosis for hemodialysis patients. J Clin Invest. 2002 Aug;110(4):437-9. doi: 10.1172/JCI16494. No abstract available. PMID 12189236
- [Derived] Marsen TA, Beer J, Mann H; German IDPN-Trial group. Intradialytic parenteral nutrition in maintenance hemodialysis patients suffering from protein-energy wasting. Results of a multicenter, open, prospective, randomized trial. Clin Nutr. 2017 Feb;36(1):107-117. doi: 10.1016/j.clnu.2015.11.016. Epub 2015 Dec 12. PMID 26708726